CLINICAL TRIAL: NCT04954859
Title: A Prospective, Multi-Centre Study (B-Sure) to Evaluate Long-Term Durability of Treatment Response in Chronic Hepatitis B Participants With and Without Nucleos(t)Ide Therapy Who Have Participated in a Previous Bepirovirsen Treatment Study
Brief Title: Long-term Follow-up Study to Evaluate Durability of Treatment Response in Previous Bepirovirsen Study Participants (B-Sure)
Acronym: B-Sure
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 206882; 2023-506867-33 (Other: EU CT Number)
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Hepatitis B
Keywords: Bepirovirsen; B-Sure; Nucleos(t)ide; Durability; HBsAg; Functional cure
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Not-on-NA participants (Experimental): Participants rolling over from study 209668 who have not received nucleos(t)ide analogue (NA) therapy during the parent study and remain off NAs will be included in this arm. Participants will be followed up for 33 months. Participants maintaining either functional cure (FC) or a partial response off NA treatment at Month 33 will be eligible to be followed up for an additional 2 years. No study treatment will be administered in this study.
  Interventions: Drug: Bepirovirsen; Drug: Placebo
- On-NA participants (Experimental): Participants rolling over from studies 209668, 209348, 212602, 202009, 219288, and 217023 who entered the parent study on stable NA therapy and remained on NA therapy for the duration of the treatment and follow-up periods in the parent study will be included in this arm. NA cessation will occur at 3 months in 206882 for eligible and willing participants. Participants will be followed up for 33 months. Participants rolling over from studies 209668 and 209348 who stopped NA treatment and are maintaining either FC or a partial response at Month 33, and remaining off NA treatment, will be eligible to be followed up for an additional 2 years. No study treatment will be administered in this study.
  Interventions: Drug: Bepirovirsen; Drug: Placebo
- NA-cessated participants (Experimental): Participants rolling over from studies 202009 and 219288 who have stopped NA treatment during the parent study will be included in this arm. Participants will be followed up for 33 months. No study treatment will be administered in this study.
  Interventions: Drug: Bepirovirsen; Drug: Placebo

INTERVENTIONS:
Drug: Bepirovirsen — No study drug will be administered in this study. Eligible participants who received prior treatment with bepirovirsen in the parent studies will be included.
Drug: Placebo — No study drug will be administered in this study. Eligible participants who received prior treatment with placebo in the parent studies (209668, 202009, and 219288) will be included to maintain the blind in the still ongoing parent studies.

SUMMARY:
This is a global multi-center, long-term follow-up study to assess durability of efficacy, as measured by maintenance of treatment response from the parent study, in participants who participated in a previous bepirovirsen study and achieved a complete or partial response. Eligible participants will be enrolled in this study after completing the end of study (EoS) visit in the respective parent bepirovirsen studies (studies B-Clear [209668: NCT04449029], B-Together [209348: NCT04676724], B-Fine [212602: NCT04544956], B-Well 1 [202009: NCT05630807], B-Well 2 [219288: NCT05630820], and TH HBV ASO-001 [217023: NCT05276297]). Participants will be categorized as Not-on-NA, NA-cessated, or On-NA based on their nucleos(t)ide analogue (NA) status in the parent study. No further treatment with bepirovirsen will be administered in this study.

ELIGIBILITY:
Inclusion criteria:

* Participants who enter the study on stable NA are willing and able to cease their NA treatment in accordance with the NA cessation schedule.
* Capable of giving informed consent.

For participants rolling over from 209668 (B-Clear), 209348 (B-Together), and 212602 (B-Fine):

* Participants who have previously received at least one dose of bepirovirsen AND

  1. Achieved the PSPO in the parent study and who maintained a response until the End of Study (EoS) visit in their parent study (defined as complete responders to bepirovirsen from the parent study) OR
  2. Demonstrated hepatitis B virus surface antigen (HBsAg) reduction greater than or equal to (≥) 1.0 log10 international units per milliliter (IU/mL) from parent study Baseline with HBsAg levels less than (<) 100 IU/mL and HBV deoxyribonucleic acid (DNA) < lower limit of quantification (LLOQ) for 24 weeks after the actual end of treatment regimen, in the absence of rescue medication and maintained until their EoS visit in the parent study.

For participants rolling over from 202009 (B-Well1) and 219288 (B-Well 2):

* Participants who have previously received at least 1 dose of bepirovirsen (or matching placebo where appropriate) AND

  1. NA cessated at Week 48 in parent study and achieved at least HBsAg <1 IU/ml and HBV DNA <LLOQ at the EOS visit (Week 96) in the parent study OR
  2. Achieved NA cessation criteria at Week 48 in parent study but have not stopped NA treatment, and are maintaining at least HBsAg <1 IU/ml and HBV DNA <LLOQ at EOS visit (Week 72) of parent study OR
  3. Did not achieve NA cessation criteria in parent study but achieved at least HBsAg <1 IU/ml and HBV DNA <LLOQ at EOS visit (Week 72) of parent study.

For participants rolling over from 217023 (TH HBV ASO-001):

* Participants who have previously received at least 1 dose of bepirovirsen AND

  1. Achieved HBsAg <1 IU/ml and HBV DNA <LLOQ in parent study at Week 66 (ASO12 arm) or Week 78 (ASO 24 arm) and are maintaining HBsAg < 1 IU/ml and HBV DNA <LLOQ, at the EOS study visit [Week 133 ASO12 arm), or Week 145 (ASO24 arm)] in parent study OR
  2. Did not achieve HBsAg <1 IU/ml and HBV DNA <LLOQ in parent study at Week 66 (ASO12 arm) or Week 78 (ASO24 arm) but have achieved HBsAg < 1 IU/ml and HBV DNA < LLOQ by the EOS visit (Week 133 (ASO12 arm) or Week 145 (ASO24 arm)) in the parent study.

Exclusion Criteria:

* Participants who have/or are currently participating in another non-GSK interventional clinical study exploring HBV treatment since completing their treatment with bepirovirsen.
* Any condition which, in the opinion of the investigator or Medical Monitor, contraindicates their participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2029-02-08 (Estimated); Study Completion 2029-02-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Not-on-NA participants without loss of parent study primary outcome (PSPO) | From primary endpoint assessment in the parent study up to Month 57
  NA indicates nucleos(t)ide analogue (NA).
Percentage of On-NA participants rolling over from studies 209668 and 209348 without loss of functional cure (FC) after NA-cessation in study 206882 | From Month 3 up to Month 57
Percentage of On-NA participants rolling over from study 217023 without loss of FC after NA-cessation in study 206882 | From Month 3 up to Month 33
Percentage of NA-cessated participants rolling over from studies 202009 and 219288 without loss of FC after NA-cessation in the parent study | From primary endpoint assessment in the parent study up to Month 33

SECONDARY OUTCOMES:
Percentage of On-NA and NA-cessated participants with PSPO in the parent study who have hepatitis B surface antigen (HBsAg) reversion or use of any rescue medication after NA cessation (in either parent study or study 206682) | Up to Month 57
Percentage of On-NA and NA-cessated participants with PSPO in the parent study who have virologic relapse or use of any rescue medication after NA cessation (in either parent study or study 206682) | Up to Month 57
Percentage of On-NA and NA-cessated participants with PSPO in the parent study who have clinical relapse or use of any rescue medication after NA cessation (in either parent study or study 206682) | Up to Month 57
Percentage of On-NA and NA-cessated participants with PSPO in the parent study who receive NA retreatment after NA cessation (in either parent study or study 206682) | Up to Month 57
Percentage of On-NA participants with PSPO in the parent study, who continue NA treatment in study 206882, and have no loss of treatment response | From primary endpoint assessment in the parent study up to Month 33
Percentage of Not-on-NA participants with a partial response in the parent study and a delayed FC in study 206882 in absence of rescue medication after end of treatment in the parent study | Up to Month 57
Time to loss of FC from time of achieving delayed FC in Not-on-NA participants with a partial response in the parent study and a delayed FC in study 206882 | From date of achieving delayed FC up to Month 57
Percentage of On-NA participants with a partial response in the parent study, who discontinue NA treatment in study 206882, and have a delayed FC in 206882 in absence of rescue medication after end of treatment in the parent study | Up to Month 57
Time to loss of FC in On-NA participants who achieve a partial response in the parent study, discontinue NA treatment in study 206882 and achieve delayed FC in 206882 | From date of achieving delayed FC up to Month 57
Percentage of On-NA participants with a partial response in the parent study, who do not discontinue NA treatment in study 206882, and have a delayed treatment response in 206882 in absence of rescue medication after end of treatment in the parent study | Up to Month 33
Time to loss of treatment response in On-NA participants who achieve a partial response in the parent study, do not discontinue NA treatment in study 206882 and have a delayed treatment response in 206882 | From date of achieving delayed treatment response up to Month 33
Percentage of On-NA participants with a partial response in the parent study, who discontinue NA treatment in study 206882, and have HBsAg loss in the absence of any rescue medication after NA cessation in 206882 | From Month 3 to Month 57
Percentage of On-NA participants with a partial response in the parent study, who discontinue NA treatment in study 206882, and have virologic relapse or use of any rescue medication after NA cessation in 206882 | From Month 3 up to Month 57
Percentage of On-NA participants with a partial response in the parent study, who discontinue NA treatment in study 206882, and have clinical relapse or use of any rescue medication after NA cessation in 206882 | From Month 3 up to Month 57
Percentage of On-NA participants with a partial response in the parent study, who discontinue NA treatment in study 206882 and have use of any rescue medication after NA cessation in 206882 | From Month 3 up to Month 57
Percentage of participants with anti-HBs (antibody to HBsAg) | Up to 57 months
Percentage of participants with anti-HBe (antibody to hepatitis B e-antigen [HBeAg]) | Up to 57 months
Absolute values for HBsAg, hepatitis B virus (HBV) deoxyribonucleic acid (DNA), HBeAg (logarithm to the base 10 [log10] international units per milliliter [IU/mL]) | Up to 57 months
Change from Baseline for HBsAg, HBV DNA, HBeAg (log10 IU/mL) | Baseline (End of Study visit in the parent study) and up to 57 months
Absolute values for hepatitis B core-related antigen (HBcrAg) (kiloUnits per milliliter [kU/mL]) | Up to 57 months
Change from Baseline for HBcrAg (kU/mL) | Baseline (End of Study visit in the parent study) and up to 57 months
Absolute values for HBV ribonucleic acid (RNA) (log10 IU/ml) | Up to 57 months
Change from Baseline for HBV RNA (log10 IU/ml) | Baseline (End of Study visit in the parent study) and up to 57 months
Percentage of participants with mutations | Up to 57 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (46):
- United States (3):
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
- GSK Investigational Site, Buenos Aires, Argentina
- Bulgaria (2):
  - GSK Investigational Site, Sliven
  - GSK Investigational Site, Sofia
- Canada (3):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Toronto, Ontario
- China (3):
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Wuhan
- France (2):
  - GSK Investigational Site, Clichy
  - GSK Investigational Site, Strasbourg
- GSK Investigational Site, Pokfulam, Hong Kong
- Italy (2):
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Modena
- Japan (7):
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Lublin, Poland
- Romania (2):
  - GSK Investigational Site, Craiova Dolj
  - GSK Investigational Site, Galati
- Russia (6):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Красноярск
- GSK Investigational Site, Singapore, Singapore
- South Africa (2):
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Johannesburg
- South Korea (4):
  - GSK Investigational Site, Ansan-si Gyenggi-do
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
- Spain (2):
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santander
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Kho Hong Hat Yai
- United Kingdom (2):
  - GSK Investigational Site, London
  - GSK Investigational Site, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.